CLINICAL TRIAL: NCT03915652
Title: Addressing Disparities in Lupus Care Through an Integrated Care Management Program (Rheum-iCMP)
Brief Title: Addressing Disparities in Lupus Care Through an Integrated Care Management Program
Acronym: Rheum-iCMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Partners HealthCare (Other)
Responsible Party: Principal Investigator, Candace Hillary Feldman, MD, Assistant Professor of Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB 2019P000638
Record Dates: First submitted 2019-03-12; First posted 2019-04-16 (Actual); Results first posted 2025-01-22 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Systemic Lupus Erythematosus
Keywords: minority health; prevention; vaccine; behavior; women's health; autoimmune; intervention; survey; QI/QA; outcomes (health services/delivery)
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Behavior

STUDY DESIGN:
Intervention Model Description: The investigators plan to newly enroll 40 lupus patients prospectively using a stepped wedge design starting first with 20 patients enrolled in Rheum-iCMP, and then with 20 additional patients enrolled 4 months later. For the second 20 patients, for the first 4 months, patients will receive educational material.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rheum iCMP Wave 1 (Experimental): 20 patients enrolled immediately in Rheum iCMP
  Interventions: Behavioral: Rheum iCMP
- Rheum iCMP Wave 2 (Experimental): 20 patients enrolled in Rheum iCMP after 4 months; will receive monthly lupus educational materials mailed to their home during the first 4 months
  Interventions: Behavioral: Rheum iCMP

INTERVENTIONS:
Behavioral: Rheum iCMP — Selected iCMP nurses will receive a 4-hour training using unique educational materials already developed by our team that specifically address lupus-related racial, ethnic and socioeconomic disparities, as well as clinical information about lupus. These iCMP nurses will then reach out to high-risk lupus patients to ensure that patients attend scheduled rheumatology appointments, fill prescriptions for lupus-specific medications, and obtain recommended lupus screening labs and preventive care.

SUMMARY:
The aim of this study is to identify lupus patients receiving care at Brigham and Women's Hospital (BWH) who are at high risk for potentially avoidable acute care utilization, inconsistent ambulatory care use, and adverse outcomes. The investigators will invite high-risk lupus patients to participate in an intensive care management program with a nurse manager, and will determine whether this program improves receipt of high quality sustained outpatient care and reduces avoidable emergency department visits and hospitalizations. The investigators will also study the social determinants that contribute to acute care use and avoidable outcomes among lupus patients using semi-structured interviews and a photovoice method.

DETAILED DESCRIPTION:
The aim of this study is to determine whether an intensive care management program for high-risk lupus patients (Rheum-iCMP, modeled after the highly successful BWH iCMP for primary care patients) reduces acute care utilization (emergency department (ED) visits, hospitalizations), improves rheumatology clinic appointment attendance, and ultimately improves quality of lupus care in this group. Selected iCMP nurses will receive a 4-hour training using unique educational materials already developed by our team that specifically address lupus-related racial, ethnic and socioeconomic disparities, as well as clinical information about lupus.

The investigators plan to identify high-risk lupus patients in the Partners' risk contract (Medicaid, Medicare and certain commercial insurances) with BWH primary care physicians (PCPs) from three sources. First, the investigators will use the BWH Lupus Registry, which is updated regularly and includes lupus patients actively receiving care at BWH. Second, the investigators will identify lupus patients via Partners electronic medical record (EMR) using our validated lupus algorithm and look specifically at those receiving primary care within the BWH system. The investigators will link both BWH Lupus Registry patients and patients meeting our algorithm to claims data through the Population Health Repository. The investigators will then identify patients with increased healthcare utilization, including ED visits and/or hospitalizations during the preceding 3 years, and who are at risk for avoidable outcomes (rheumatology appointment no-shows/same-day cancellations within the same period). The investigators will also apply the Partners' Center for Population Health high-risk algorithm to both cohorts to identify additional high-risk patients. The investigators will then reach out to the identified patients' PCPs or their rheumatologists for approval to send a study invitation to patients or asking physicians to introduce the study to their patients with a fact sheet. Third, the investigators will ask rheumatologists to refer lupus patients who might benefit from Rheum-iCMP, since a similar referral system has been successful within BWH-wide iCMP.

The investigators plan to newly enroll 40 lupus patients aged ≥18 years old, both male and female, English-speaking, and who receive their primary care at BWH prospectively using a stepped wedge design starting first with 20 patients enrolled in Rheum-iCMP, and then with 20 additional patients enrolled 4 months later. For the second 20 patients, for the first 4 months, patients will receive educational material about lupus on a monthly basis. The investigators will invite these 40 patients to also participate in a semi-structured interview that includes asking participants ahead of time to take 10-15 photographs (with a disposable camera the investigators will provide) of their neighborhoods and homes, in order to begin a conversation about the social determinants that contribute to their care-seeking behaviors. Participants will then sit with a moderator for a ~60-90 minute semi-structured, in-depth photo-elicitation interview. Participants will be asked to 1) select the photographs for discussion, 2) contextualize each image and tell a story, 3) describe what is really happening and how it relates to their life and 4) propose suggestions for what can be done to improve any barriers described. The elicitation interviews will be audio-recorded, transcribed verbatim, and entered into Dedoose for analysis. Participation in the photographs/interview is not a requirement of being a part of Rheum-iCMP.

In addition to these 40 newly enrolled patients, the investigators expect that 100 additional adult lupus patients within the Partners system are already enrolled in BWH iCMP. Among these patients, the investigators plan to examine EMR and claims data pre and post iCMP enrollment as an observational study looking at differences in utilization. However, the investigators do not plan to ask for survey completion for this population since this iCMP program is considered standard of care and these patients are already a part of it. Because the investigators do not feel that this will involve more than minimal risk and because it would not be feasible, the investigators do not plan to consent these individuals to allow us to examine their medical records.

The investigators will compare lupus-related quality metrics, rheumatology appointment attendance, and acute care use 12 months after enrollment in rheum-iCMP as compared to 12 months before enrollment in rheum-iCMP. The investigators will collect surveys at 12 months after enrollment in rheum-iCMP. For individuals who unenrolled before the end of the 12-month study period, we will stop the chart review at the date of unenrollment. The investigators will also examine EMR and claims data when available prior to the rheum-iCMP and then for the subsequent 12-24 months during and following rheum-iCMP. For the lupus patients who are already enrolled in BWH iCMP, the investigators will separately compare measures extractable from EMRs and claims pre-iCMP, during iCMP but pre-lupus-specific iCMP nurse training, and during Rheum-iCMP (post- nurse training) for N=100. These data are observational/non-experimental and distinct from the pilot trial intervention and thus cannot be combined and will be analyzed separately.

During the intervention period, our project coordinator will set up a sustainable EPIC system for tracking appointment no-shows and SLE quality metrics (e.g. lab monitoring, contraceptive use). The investigators will collect the following surveys: medication adherence and medication beliefs using the MASRI survey and the Beliefs about Medications scale, lupus disease activity using SLAQ, mental health using the MHI-5, social determinants of health using the Partners Healthcare Social Determinants of Health (SDH) Survey, global health assessment using the PROMIS global health scale short form, and racial discrimination using the Everyday Discrimination Scale. The investigators will also collect baseline demographics information via a demographics survey. The investigators will determine acute care utilization (e.g. ED visits, hospitalizations) using partners risk contract claims data. The investigators will also use surveys at 12 months after rheum-iCMP enrollment to assess patient, iCMP nurse, and MD satisfaction. Surveys will be collected at outpatient appointments or via mail. For longer term quality metrics 12-24 months past the intervention period, the investigators will work with the Center for Population Health's team to set up a tracking system that has Partners-wide claims data linked with EMRs. For the 100 patients already enrolled in the iCMP intervention, the investigators assess changes in acute care use (ED visits and hospitalizations) and appointment no shows however this is an observational separate study and will not be compared to data from the newly enrolled patients. The investigators will also collect these data for the 40 newly enrolled patients, which will be analyzed separately as the intervention is different.

This is a pilot study. One of our primary measures is to reduce ambulatory rheumatology care no-show rates for the highest risk patients. The investigators estimate that the no-show rate is about 70% and the aim of this study is to reduce this rate to 20%. The investigators would need a total of 40 patients (20 in each arm) to have 80% power to detect this difference, which is why the target enrollment for new patients in Rheum-iCMP is 40.

ELIGIBILITY:
Inclusion Criteria

* Meet at least 4 American College of Rheumatology criteria for systemic lupus erythematosus (SLE) or rheumatologist diagnosis of SLE
* Over the preceding 3 years, at least 1 hospitalization or ED visit related to lupus OR at least 1 rheumatology appointment no-show or same-day cancellation
* Receive their primary care at BWH

Exclusion Criteria:

* Non-English or Spanish speaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2019-06-21 (Actual); Primary Completion 2022-07-20 (Actual); Study Completion 2025-07-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Candace H Feldman, MD, ScD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The goal enrollment in this trial was 40 individuals, and of this total, the starting N was 35. We experienced difficulties recruiting our target number of 40 individuals and exceeded the time and funding allocated to this study and thus ended enrollment after 35.
Period: Overall Study
Arm/Group | Rheum iCMP Wave 1 | Rheum iCMP Wave 2
Started | 18 | 17
Completed | 17 | 12
Not Completed | 1 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rheum iCMP Wave 1 | Rheum iCMP Wave 2 | Total
Number analyzed (Participants) | 18 | 17 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (17.5) | 47.6 (19.3) | 46.2 (18.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 30
  Male | 3 | 2 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 7 | 9
  Not Hispanic or Latino | 16 | 10 | 26
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 5 | 13
  White | 5 | 4 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 7 | 10
Region of Enrollment [Number; unit: participants]
  United States | 18 | 17 | 35
Baseline Period Appointment No Shows [Mean (Standard Deviation); unit: Appointment No Shows] — Determined 12 months prior to enrollment. Population: Participants withdrew prior to assessment of baseline outcome data.
  Appointment No Shows
    number analyzed (Participants) | 17 | 12 | 29
    (all) | 6 (9) | 8 (7) | 7 (8)
Baseline Period Acute Care Use [Mean (Standard Deviation); unit: Acute Care Visits] — Determined 12 months prior to enrollment. Population: Participants withdrew prior to assessment of baseline outcome data.
  Acute Care Visits
    number analyzed (Participants) | 17 | 12 | 29
    (all) | 1.53 (1.66) | 1.67 (2.10) | 1.59 (1.82)
Quality of Lupus Care: SLE Quality Metric Scoring System for Adults [Mean (Standard Deviation); unit: units on a scale] — SLE Quality Metric Scoring System for Adults. This includes 37 questions assessing general SLE preventive care, immunizations, cancer screening, infectious screening prior to initiation of immunosuppression, screening for cardiovascular disease, laboratory monitoring for SLE disease activity and renal involvement, reducing morbidity due to medications, reproductive health, and management of comorbid antiphospholipid syndrome. At baseline, this is the number of metrics not completed. The total score range is 0-37; higher scores mean more incomplete metrics (e.g., vaccinations not given). Population: Participants withdrew prior to assessment of baseline checklist
  units on a scale
    number analyzed (Participants) | 16 | 12 | 28
    (all) | 5.1 (1.89) | 5.75 (2.67) | 5.39 (2.23)
Medication Adherence Self-Report Inventory (MASRI) [Mean (Standard Deviation); unit: units on a scale] — This is a medication adherence scale, scored based on an individual's indication on a VAS (0 to 100) of their degree of medication adherence. Population: Subset of the population returned completed baseline and follow-up surveys.
  units on a scale
    number analyzed (Participants) | 2 | 4 | 6
    (all) | 90 (0) | 97.5 (5) | 95 (5.5)
Beliefs about Medications Survey [Mean (Standard Deviation); unit: units on a scale] — Population: All participants did not complete baseline and follow-up surveys for secondary outcomes.
  units on a scale
    number analyzed (Participants) | 3 | 4 | 7
    (all) | 2.53 (0.81) | 2.4 (1.01) | 2.46 (0.85)
Lupus Disease Activity (SLAQ) [Mean (Standard Deviation); unit: units on a scale] — Population: All participants did not complete baseline and follow-up surveys for secondary outcomes.
  units on a scale
    number analyzed (Participants) | 2 | 3 | 5
    (all) | 10 (7.07) | 16.3 (13.8) | 15.5 (8.23)
Depressive Symptoms Scale (MHI-5) [Mean (Standard Deviation); unit: units on a scale] — Population: All participants did not complete baseline and follow-up surveys for secondary outcomes.
  units on a scale
    number analyzed (Participants) | 2 | 2 | 4
    (all) | 48 (22.6) | 62 (19.8) | 55 (19.1)
PROMIS Patient Reported Global Health - Physical Health [Mean (Standard Deviation); unit: units on a scale] — Population: All participants did not complete baseline and follow-up surveys for secondary outcomes.
  units on a scale
    number analyzed (Participants) | 3 | 3 | 6
    (all) | 43.2 (2.94) | 43.2 (1.50) | 43.2 (2.09)
Social Determinants of Health (SDoH) Number of Needs [Mean (Standard Deviation); unit: units on a scale] — Indication of the number of social determinants of health-related needs (e.g., food insecurity, housing instability) on a survey asking about presence or absence of these needs. The range was 0-8; higher scores indicate more needs. Population: All participants did not complete baseline and follow-up surveys for secondary outcomes.
  units on a scale
    number analyzed (Participants) | 3 | 4 | 7
    (all) | 1.67 (1.15) | 1.25 (0.96) | 1.43 (0.98)
Everyday Discrimination Scale [Mean (Standard Deviation); unit: units on a scale] — A measure of experiences of discrimination. Population: All participants did not complete baseline and follow-up surveys for secondary outcomes.
  units on a scale
    number analyzed (Participants) | 3 | 4 | 7
    (all) | 8 (7.55) | 0.5 (1) | 3.71 (5.96)

OUTCOME MEASURES:

1. Primary Outcome: Lupus-related Appointment Nonadherence
Description: Mean change in the number of lupus-related ambulatory care visit no-shows and same-day cancellations
Time Frame: Mean change from 12 months prior to intervention and the 12 months during the intervention
Measure: Mean (Standard Deviation); unit: Appointment No Shows
Arm/Group | Rheum iCMP Wave 1 | Rheum iCMP Wave 2
Number analyzed (Participants) | 17 | 12
Appointment No Shows | 6.2 (7.4) | 5.2 (5.6)
Statistical Analysis 1: Comparison: Rheum iCMP Wave 1 vs Rheum iCMP Wave 2; Waves 1 and 2 were combined and appointment nonadherence during the intervention was compared with the 12 months prior; Test type: Superiority; p = 0.34, t-test, 2 sided; Paired t-test; Mean Difference (Final Values) = -0.93, 95% CI 2-sided [-2.88 to 1.02]

2. Primary Outcome: Composite Measure of Acute Care Utilization
Description: Mean change in the number of ED visits plus number of hospitalizations
Time Frame: Mean change from 12 months prior to intervention and the 12 months during the intervention
Measure: Mean (Standard Deviation); unit: Acute Care Use Visits
Arm/Group | Rheum iCMP Wave 1 | Rheum iCMP Wave 2
Number analyzed (Participants) | 17 | 12
Acute Care Use Visits | 1.29 (2.54) | 1.17 (1.90)
Statistical Analysis 1: Comparison: Rheum iCMP Wave 1 vs Rheum iCMP Wave 2; Waves 1 and 2 were combined and emergency department visits and hospitalizations during the intervention was compared with the 12 months prior; Test type: Superiority; p = 0.34, t-test, 2 sided; Paired t-test; Mean Difference (Final Values) = -0.34, 95% CI 2-sided [-1.08 to 0.39]

3. Primary Outcome: Quality of Lupus Care: SLE Quality Metric Scoring System for Adults
Description: Percent of quality metrics from the SLE Quality Metric Scoring System for Adults remaining from baseline 12 months after the start of the intervention. The percent of needs remaining at 12 months was determined and the mean (SD) percent of remaining needs was calculated by arm. Percentages can range from 0-100, with 100 meaning that more quality metrics were not completed (worse outcome).
Time Frame: Percent of quality metrics remaining at 12 months
Measure: Mean (Standard Deviation); unit: Percent of score
Arm/Group | Rheum iCMP Wave 1 | Rheum iCMP Wave 2
Number analyzed (Participants) | 17 | 12
Percent of score | 64 (32) | 53 (41)
Statistical Analysis 1: Comparison: Rheum iCMP Wave 1 vs Rheum iCMP Wave 2; Wave 1 and Wave 2 were combined and the quality metric at the end of the 12-month intervention was compared to the metric from the start of the intervention; Test type: Superiority; p < 0.001, t-test, 1 sided; One sided t-test of percent of needs remaining from 100%; Mean Difference (Final Values) = 0.59, 95% CI 2-sided [0.45 to 0.73]

4. Secondary Outcome: Medication Adherence Self-Report Inventory (MASRI)
Description: Mean change in MASRI score (for lupus medications) from baseline to 12 months. Score range is 0-100. Higher scores indicate greater adherence (on a scale from 0 to 100, 100 indicating a person's rating of perfect adherence).
Time Frame: Mean change from baseline to 12 months after the start of the intervention.
Population: Subset of the population who returned completed baseline and follow-up surveys.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rheum iCMP Wave 1 | Rheum iCMP Wave 2
Number analyzed (Participants) | 2 | 4
units on a scale | 65 (49.5) | 98.8 (2.5)
Statistical Analysis 1: Comparison: Rheum iCMP Wave 1 vs Rheum iCMP Wave 2; Test type: Superiority; p = 0.51, t-test, 2 sided; Mean Difference (Final Values) = 7.5, 95% CI 2-sided [-19.8 to 34.8]

5. Secondary Outcome: Beliefs About Medications Survey
Description: Mean change in Beliefs About Medications score (for lupus medications) from baseline to 12 months after the start of the intervention. Score range is 5-25. Higher scores indicate a worse outcome (higher scores indicate more negative feelings about lupus medications).
Time Frame: Mean change from baseline compared to 12 months after the start of the intervention
Population: Participants who completed baseline and follow-up surveys.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rheum iCMP Wave 1 | Rheum iCMP Wave 2
Number analyzed (Participants) | 3 | 4
units on a scale | 2.13 (1.14) | 1.4 (0.43)
Statistical Analysis 1: Comparison: Rheum iCMP Wave 1 vs Rheum iCMP Wave 2; Waves 1 and 2 combined, compared post to pre; Test type: Superiority; p = 0.17, t-test, 2 sided; Paired t-test; Mean Difference (Final Values) = 0.74, 95% CI 2-sided [-0.43 to 1.92]

6. Secondary Outcome: Systemic Lupus Activity Questionnaire (SLAQ)
Description: Mean change in patient-reported lupus disease activity from baseline to 12 months using the SLAQ score. Score range is 0-46. Higher scores indicate a worse outcome (higher scores indicate more lupus disease activity).
Time Frame: Mean change from baseline compared to 12 months after the start of the intervention
Population: Individuals who completed baseline and follow-up surveys
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rheum iCMP Wave 1 | Rheum iCMP Wave 2
Number analyzed (Participants) | 2 | 3
units on a scale | 11 (7.07) | 14.3 (4.93)
Statistical Analysis 1: Comparison: Rheum iCMP Wave 1 vs Rheum iCMP Wave 2; Waves 1 and 2 combined, compared pre/post intervention; Test type: Superiority; p = 0.72, t-test, 2 sided; Paired t-test; Mean Difference (Final Values) = 0.8, 95% CI 2-sided [-4.92 to 6.52]

7. Secondary Outcome: Mental Health Inventory-5 (MHI-5)
Description: Mean change in depressive or anxious symptoms from baseline to 12 months using the MHI-5 survey. Score range is 0-100. Higher scores indicate a better outcome (higher scores indicate better mental health).
Time Frame: Mean change from baseline compared to 12 months after the start of the intervention
Population: Participants who completed baseline and follow-up surveys
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rheum iCMP Wave 1 | Rheum iCMP Wave 2
Number analyzed (Participants) | 2 | 2
units on a scale | 48 (17) | 58 (14.1)
Statistical Analysis 1: Comparison: Rheum iCMP Wave 1 vs Rheum iCMP Wave 2; Waves 1 and 2 are combined; pre/post survey analysis; Test type: Superiority; p = 0.50, t-test, 2 sided; Mean Difference (Final Values) = 2, 95% CI 2-sided [-6.22 to 10.22]

8. Secondary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS) Global Health Scale Short Form
Description: Mean change in global health from baseline to 12 months using the PROMIS global health scale short form. Score range is 9-45. Higher scores indicate a better outcome (higher scores indicate improved global health and well-being).
Time Frame: Mean change from baseline compared to 12 months after the start of the intervention
Population: Participants who completed baseline and follow-up surveys.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rheum iCMP Wave 1 | Rheum iCMP Wave 2
Number analyzed (Participants) | 3 | 3
units on a scale | 39 (2.76) | 39.8 (4.27)
Statistical Analysis 1: Comparison: Rheum iCMP Wave 1 vs Rheum iCMP Wave 2; Waves 1 and 2 combined; pre/post analysis; Test type: Superiority; p = 0.01, t-test, 2 sided; Mean Difference (Final Values) = 3.77, 95% CI 2-sided [1.06 to 6.47]

9. Secondary Outcome: Social Determinants of Health (SDOH) Survey
Description: Percent of social determinants of health (SDoH)-related needs at 12 months from baseline using the SDoH Survey. The survey range is 0-8 and the percent of remaining needs is 0-100 with 100 meaning that all of the needs remain (worse outcome).
Time Frame: Percent of social determinants of health-related needs remaining 12 months after the start of the intervention
Population: Participants who completed baseline and follow-up surveys.
Measure: Mean (Standard Deviation); unit: Percent of baseline score
Arm/Group | Rheum iCMP Wave 1 | Rheum iCMP Wave 2
Number analyzed (Participants) | 3 | 4
Percent of baseline score | 2.33 (1.15) | 1 (1.41)
Statistical Analysis 1: Comparison: Rheum iCMP Wave 1 vs Rheum iCMP Wave 2; Waves 1 and 2 combined, pre/post test; Test type: Superiority; p = 0.77, t-test, 2 sided; Paired t-test; Mean Difference (Final Values) = -0.14, 95% CI 2-sided [-1.27 to 0.98]

10. Secondary Outcome: Everyday Discrimination Scale
Description: Mean change in daily discrimination encountered from baseline to 12 months using the Everyday Discrimination Scale. Score range is 0-40. Higher scores indicate a worse outcome (higher scores indicate a greater amount of discrimination encountered).
Time Frame: Mean change from baseline compared to 12 months after the start of the intervention
Population: Participants who completed baseline and follow-up surveys.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rheum iCMP Wave 1 | Rheum iCMP Wave 2
Number analyzed (Participants) | 3 | 4
units on a scale | 1.33 (1.15) | 1.75 (2.87)
Statistical Analysis 1: Comparison: Rheum iCMP Wave 1 vs Rheum iCMP Wave 2; Waves 1 and 2 combined; pre/post analysis; Test type: Superiority; p = 0.37, t-test, 2 sided; Paired t-test; Mean Difference (Final Values) = 2.14, 95% CI 2-sided [-3.23 to 7.52]

ADVERSE EVENTS:
Time Frame: 1 year study period
Description: Hospitalizations and emergency department visits were not considered adverse events as they were primary outcome measures for this study and thus are reported as such. No adverse events occurred during the time course of this study and thus the educational component and the intervention component were combined in this report.
Arm/Group | Rheum iCMP Wave 1 | Rheum iCMP Wave 2
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/17
Other Adverse Events (participants affected / at risk) | 0/18 | 0/17

LIMITATIONS AND CAVEATS:
A small percentage of participants returned their baseline and follow-up surveys which will limit interpretability of secondary outcome data. Primary outcomes came from chart review data and therefore this is complete and interpretable for the participants who did not withdraw.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-27): https://cdn.clinicaltrials.gov/large-docs/52/NCT03915652/Prot_SAP_000.pdf